CLINICAL TRIAL: NCT01078909
Title: Dose Response Effects of Marine Omega-3 Fatty Acids on Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKE LPS
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease; Inflammation
Keywords: Cardiovascular disease; Inflammation; Fish Oil; Omega-3 Fatty Acids; LPS; Endotoxin
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 300mg Fish Oil (EPA + DHA) Supplement (Experimental)
  Interventions: Biological: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA)
- 600mg Fish Oil (EPA+DHA) Supplement (Experimental)
  Interventions: Biological: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA)
- 900mg Fish Oil (EPA + DHA) Supplement (Experimental)
  Interventions: Biological: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA)
- 1800mg Fish Oil (EPA + DHA) Supplement (Experimental)
  Interventions: Biological: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA)
- Placebo (Placebo Comparator)
  Interventions: Biological: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA)

INTERVENTIONS:
Biological: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA) — Comparison of 4 doses of EPA+DHA on in vivo and ex vivo (monocytes) response to an inflammatory stimulus (endotoxin) following a 6 month supplementation period
  Other Names: Omega-3 Fatty Acids; Fish Oil

SUMMARY:
The purpose of this study is to determine the lowest effective dose of EPA + DHA (300, 600, 900 and 1,800 mg/day delivered as fish oil supplements) that significantly attenuates the inflammatory response to in vivo and ex vivo endotoxin challenge as measured by the production over time of several inflammatory markers.

DETAILED DESCRIPTION:
Inflammation is an important biological process initiated by the immune system in response to injury, irritation or infection. Prolonged or chronic inflammation is involved in the etiology of several diseases such as cardiovascular disease (CVD), diabetes, rheumatoid arthritis, cancer, and neurodegenerative diseases such as Alzheimer disease. The evidence base clearly demonstrates benefits of diet in ameliorating inflammation and reducing the burden of chronic disease. With respect to marine-derived omega-3 fatty acids and various markers of inflammation related to cardiovascular disease (CVD), both population studies and randomized controlled supplementation trials have yielded mixed results.

Some studies have demonstrated a dose-response relationship between dietary eicosapentaenoic acid and docosahexaenoic acid (EPA + DHA) and increased membrane (phospholipid) EPA and DHA. Red blood cell (RBC) EPA + DHA content has been proposed as a potential, modifiable marker for coronary heart disease (CHD) risk. It is well established that these fatty acids are precursors of series-3 prostanoids, thromboxanes, 5-series leukotrienes, and novel lipid mediators such as resolvins and protectins that have anti-inflammatory effects. We hypothesize that nutritionally-relevant intakes of omega-3 fatty acids are able to blunt the usual response to an inflammatory stimulus. We propose to test this hypothesis using both in vivo (i.v. endotoxin challenge) and ex vivo (endotoxin-stimulated monocytes) models in a 6-month, dose-response study with marine-derived omega-3 fatty acid supplements in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant/lactating women between the ages of 20 and 45
* BMI >19.9 and <30.0
* Able to give written informed consent and willing to comply with all study- related procedures.

Exclusion Criteria:

* Previous history of heart disease or diabetes
* Renal Insufficiency
* Chronic anti-inflammatory use
* Systolic blood pressure < 90
* Individuals currently using tobacco products or have done so in the previous 30 days
* Individuals taking Omega-3 fatty acid supplements or their usual intake of fish is greater than 3-4 servings per month.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon L Jensen, MD, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Flock MR, Skulas-Ray AC, Harris WS, Etherton TD, Fleming JA, Kris-Etherton PM. Determinants of erythrocyte omega-3 fatty acid content in response to fish oil supplementation: a dose-response randomized controlled trial. J Am Heart Assoc. 2013 Nov 19;2(6):e000513. doi: 10.1161/JAHA.113.000513. PMID 24252845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and screened occured between September 2011 and March 2012 at the Clinical Research Center at Penn State University.
Pre-assignment Details: A computer-generated randomization scheme was developed in advance. The randomization scheme was stratified by sex and age and used a balanced block size of 5 to ensure even distribution among treatment groups. Using this randomization scheme, eligible participants were assigned to blinded treatments at the baseline visit by the study coordinator.
Groups:
- 300mg Fish Oil (EPA + DHA) Supplement; 600mg Fish Oil (EPA+DHA) Supplement; 900mg Fish Oil (EPA + DHA) Supplement; 1800mg Fish Oil (EPA + DHA) Supplement; Placebo: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA) following a 6 month supplementation period
Period: Overall Study
Arm/Group | 300mg Fish Oil (EPA + DHA) Supplement | 600mg Fish Oil (EPA+DHA) Supplement | 900mg Fish Oil (EPA + DHA) Supplement | 1800mg Fish Oil (EPA + DHA) Supplement | Placebo
Started | 25 | 25 | 25 | 25 | 25
Completed | 23 | 21 | 24 | 24 | 23
Not Completed | 2 | 4 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- 300mg Fish Oil (EPA + DHA) Supplement; 600mg Fish Oil (EPA+DHA) Supplement; 1800mg Fish Oil (EPA + DHA) Supplement; Placebo: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA) following a 5 month supplementation period
- 900mg Fish Oil (EPA + DHA) Supplement: Eicosapentaenoic Acid and Docosahexaenoic Acid (EPA + DHA) following a 65 month supplementation period
- Total: Total of all reporting groups
Arm/Group | 300mg Fish Oil (EPA + DHA) Supplement | 600mg Fish Oil (EPA+DHA) Supplement | 900mg Fish Oil (EPA + DHA) Supplement | 1800mg Fish Oil (EPA + DHA) Supplement | Placebo | Total
Number analyzed (Participants) | 23 | 21 | 24 | 24 | 23 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (7.2) | 27.1 (7.3) | 25.8 (6.4) | 26.0 (5.9) | 25.7 (6.7) | 26.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 11 | 11 | 12 | 55
  Male | 12 | 11 | 13 | 13 | 11 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Concentrations of Inflammatory Markers (TNF-alpha and IL-6) Following 5 Months of Treatment
Time Frame: 5 months
Population: One individual was removed from the analysis due to having very high RBC EPA+DHA content at study entry (>8%)
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | 300mg Fish Oil (EPA + DHA) Supplement | 600mg Fish Oil (EPA+DHA) Supplement | 900mg Fish Oil (EPA + DHA) Supplement | 1800mg Fish Oil (EPA + DHA) Supplement | Placebo
Number analyzed (Participants) | 23 | 21 | 24 | 23 | 23
pg/mL
  TNF-alpha (pg/mL) | 1.4 [1.3 to 1.5] | 1.3 [1.1 to 1.5] | 1.4 [1.2 to 1.5] | 1.5 [1.2 to 1.6] | 1.4 [1.1 to 1.6]
  IL-6 (pg/mL) | 0.9 [0.7 to 1.1] | 1 [0.8 to 1.2] | 0.9 [0.7 to 1.1] | 1 [0.8 to 1.2] | 0.9 [0.7 to 1.1]

2. Primary Outcome: Mean Concentrations of CRP Following 5 Months of Treatment
Time Frame: 5 months
Population: One individual was removed from the analysis due to having very high RBC EPA+DHA content at study entry (>8%)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 300mg Fish Oil (EPA + DHA) Supplement | 600mg Fish Oil (EPA+DHA) Supplement | 900mg Fish Oil (EPA + DHA) Supplement | 1800mg Fish Oil (EPA + DHA) Supplement | Placebo
Number analyzed (Participants) | 23 | 21 | 24 | 23 | 23
mg/dL | 0.6 [0.4 to 1.1] | 0.5 [0.3 to 0.6] | 0.6 [0.4 to 1.0] | 0.6 [0.4 to 0.9] | 0.5 [0.3 to 0.8]

3. Secondary Outcome: Change in Lipid Mediators
Description: 0 Participants Analyzed; Lipid mediators were unable to be detected therefore there are no data to report.
Time Frame: 1, 2, 3 and 5 days post LPS administration
Population: Lipid mediators were unable to be detected; Data were not collected.
Arm/Group | 300mg Fish Oil (EPA + DHA) Supplement | 600mg Fish Oil (EPA+DHA) Supplement | 900mg Fish Oil (EPA + DHA) Supplement | 1800mg Fish Oil (EPA + DHA) Supplement | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 300 mg/d EPA + DHA (Fish Oil) Supplement | 600 mg/d EPA + DHA (Fish Oil) Supplement | 900 mg/d EPA + DHA (Fish Oil) Supplement | 1800 mg/d EPA + DHA (Fish Oil) Supplement | 0 mg/d EPA + DHA (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/24 | 0/24 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes